CLINICAL TRIAL: NCT04198090
Title: Efficacy of Sexual & Gender Minority Competency in Oncology Practice
Brief Title: Sexual & Gender Minority Competency in Oncology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Principal Investigator, Charles Kamen, Assistant Professor, University of Rochester
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: UCC19177
Record Dates: First submitted 2019-12-10; First posted 2019-12-13 (Actual); Last update posted 2022-01-14 (Actual); Status verified 2022-01

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: Single-arm, open-label trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Sexual & Gender Minority (SGM) Competence Training (Other): Personnel will be trained using a validated, two-hour long SGM curriculum created by the Fenway Institute and tailored for Oncology.
  Interventions: Behavioral: SGM Competency Training Program

INTERVENTIONS:
Behavioral: SGM Competency Training Program — A validated, two-hour long SGM curriculum created by the Fenway Institute and tailored for oncology

SUMMARY:
This study is a single-arm, open-label trial of a sexual and gender minority (SGM) competence training program at Wilmot Cancer Institute (Wilmot) and its regional care locations (e.g., Wilmot Medical Oncology, Wilmot Radiation Oncology, Gynecological Oncology, Highland Hospital, Pluta Cancer Center). Results will be descriptive in nature and will be used to inform a R01 grant application.

The investigators will train Wilmot personnel (physicians, nurses, other providers, staff, and administrators) at each care location using a validated, two-hour long SGM curriculum created by the Fenway Institute and tailored for oncology. The investigators will collect data from all personnel on knowledge and attitudes about SGM patients before and after the training. After the training is complete, the investigators will recruit 5 SGM patients and 5 heterosexual/cisgender (H/C) patients from each care location to provide data on their satisfaction with care, outcomes, and experiences.

DETAILED DESCRIPTION:
This study is a single-arm, open-label trial of a sexual and gender minority (SGM) competence training program at Wilmot Cancer Institute (Wilmot) and its regional care locations (e.g., Wilmot Medical Oncology, Wilmot Radiation Oncology, Gynecological Oncology, Highland Hospital, Pluta Cancer Center). Results will be descriptive in nature and will be used to inform a R01 grant application.

The investigators will train Wilmot personnel (physicians, nurses, other providers, staff, and administrators) at each care location using a validated, two-hour long SGM curriculum created by the Fenway Institute and tailored for oncology. The investigators will collect data from all personnel on knowledge and attitudes about SGM patients before and after the training. Because competent communication may manifest in subtle, automatic, non-verbal processes, the investigators will also video record and analyze clinical interactions between SGM patients, heterosexual/cisgender (H/C) patients, and their oncologists. This study has four aims:

Aim 1: To test whether a SGM competence intervention improves knowledge and attitudes among Wilmot personnel (on a 8 item questionnaire) from pre- to post-training.

Aim 2: To explore patient satisfaction (on the Hospital Consumer Assessment of Healthcare Providers and Systems, HCAHPS) in Wilmot care locations both before and after our SGM competence intervention.

Aim 3: To explore patient stress (psychological distress on the Brief Symptom Inventory, anticipatory stigma on the Expectations of Rejection Scale, and experiences of discrimination on the Everyday Discrimination Scale) before and after a SGM competence intervention.

Aim 4: To explore non-verbal synchrony by conducting Motion Energy Analysis (MEA) in video recordings of clinical discussions between SGM cancer patients and their oncologists vs. H/C cancer patients and their oncologists.

ELIGIBILITY:
We will train cancer care personnel using our in-person SGM competency training.

Personnel must:

1. be a provider (physician, nurse, etc.), staff member, or administrator employed at a Wilmot care location;
2. be age 18 or older;
3. be able to understand English or American Sign Language (ASL, as training will be conducted in English with an ASL interpreter) and read English (as measures will be in English);
4. provide written informed consent.

Patients must:

1. have been diagnosed with any type of cancer;
2. be scheduled for an oncology-related visit (before, during, or after cancer treatment) at a Wilmot care location;
3. identify as a sexual and/or gender minority (SGM; e.g., preferring to partner with individuals of the same gender, identifying as a gender that differs from sex assigned at birth) or heterosexual and cisgender (H/C, for the comparison group; i.e., preferring to partner with individuals of the opposite gender and identifying as a gender that matches sex assigned at birth);
4. be age 18 or older;
5. be able to read and understand English (as measures and interviews will be in English);
6. provide written informed consent.

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients must identify as a sexual and/or gender minority (SGM; e.g., preferring to partner with individuals of the same gender, identifying as a gender that differs from sex assigned at birth) or heterosexual and cisgender (H/C, for the comparison group; i.e., preferring to partner with individuals of the opposite gender and identifying as a gender that matches sex assigned at birth)
Enrollment: 62 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Testing SGM competence | Pre- to post-training
  Personnel outcomes pre and post training will be measured using an 8-item tool created by the Fenway Institute. This tool measures knowledge about disparities and needs of SGM cancer patients, as well as attitudes about treating SGM patients. Items are rated on a 4-point scale and summed to create an overall score ranging from 0 to 32; higher scores signify better knowledge and attitudes.
Exploring Patient Satisfaction | Cross-sectional over 1 year
  Patient satisfaction with care will be measured by the Hospital Consumer Assessment of Healthcare Providers and Systems (HCAHPS, 9 items).82 HCAHPS is a national, standard, publicly reported survey of patients' perspectives on healthcare. Items measure perceived physician understanding of patient goals and communication about healthcare choices, as well as an overall rating of care received. Items can be averaged into a composite score ranging from 0 to 5, with 4-5 indicating high satisfaction.
Exploring Patient Stress | Cross-sectional over 1 year
  Psychological distress will be measured with the Brief Symptom Inventory (BSI-18).83,84 The BSI is an 18-item measure with three 6-item somatization, anxiety, and depression scales, as well as a total score (our outcome). The BSI has been well-validated in multiple studies as a measure of psychological distress in patients with various medical illnesses,85 including cancer.86 The BSI served as a convergent validity measure in developing the Distress Thermometer now recommended by the National Comprehensive Cancer Network for screening cancer patients for distress.87 Items are rated on a 4-point scale, summed, and the total score is converted to a standardized T-score; higher scores indicate higher distress.
Exploring perspectives of SGM patients | Cross-sectional over 1 year
  We will video record clinical interactions between 5 SGM cancer patients and their oncologists, as well as 5 H/C cancer patients and their oncologists. All analyses will be performed with Motion Energy Analysis (MEA) to obtain an overall estimate of nonverbal synchrony.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Kamen, PhD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

IPD SHARING:
Plan to Share IPD: No